CLINICAL TRIAL: NCT04943588
Title: Treating Hepatitis C in Pakistan. Strategies to Avoid Resistance to Antiviral Drugs
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Aga Khan University (Other); Dow University of Health Sciences (Other); University of Oxford (Other); University of Bristol (Other)
Responsible Party: Principal Investigator, Naheed Choudhry, Senior Project Manager, Queen Mary University of London
Other Study IDs: PakHepCscreen
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — We will take Blood samples to test presence of Hepatitis C RNA only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HCV Negative: At initial screen, this population will be HCV negative via the diagnostic testing. They will be eligible if they fulfil the following:
  1. over 18 yrs old.
  2. willing to participate
  3. no previous history of therapy with oral medication for chronic HCV infection
  Interventions: Diagnostic Test: HCV Antibody test (Point of care)
- HCV Positive with first-line treatment success: At the initial screen, this population (approx. 5000) will be HCV RNA positive and will undergo 12/24 week treatment of sofosbuvir plus daclatasvir. After treatment, their blood sample will show that they have achieved a sustained virological response (SVR) defined as HCV RNA undetectable.
  Interventions: Diagnostic Test: HCV RNA (PCR)
- HCV positive with first-line treatment failure: At the initial screen, this population (approx. 5000) will be HCV RNA positive and will undergo 12/24 week treatment of sofosbuvir/daclatasvir. After treatment, this proportion of people will NOT achieve an (SVR - defined as HCV RNA undetectable).
  Interventions: Diagnostic Test: HCV RNA (PCR)
- Cirrhotic Patients: Hepatitis C RNA positive that have cirrhosis
  Interventions: Diagnostic Test: AST/ALT and platelets measurement

INTERVENTIONS:
Diagnostic Test: HCV RNA (PCR) — We will test HCV positive patients after treatment to observe if they achieve SVR
  Groups: HCV Positive with first-line treatment success; HCV positive with first-line treatment failure
Diagnostic Test: HCV Antibody test (Point of care) — HCV antibody test used to establish if patients have had or are actively infected with HCV
  Groups: HCV Negative
Diagnostic Test: AST/ALT and platelets measurement — AST/ALT and platelets to determine APRI score
  Groups: Cirrhotic Patients

SUMMARY:
We will determine how best to manage the hepatitis C virus (HCV) epidemic in Pakistan by measuring effectiveness of Pakistan-government sponsored current therapies, emergence of viral resistance, consequences of infection (chiefly liver cancer) and through developing models, based on incidence data, determine the proportion of people who need curative treatment to eliminate HCV, and assess whether targeting can optimise this.

DETAILED DESCRIPTION:
Chronic infection with the hepatitis C virus (HCV) causes liver damage and, in many, liver cancer. We have effective drugs allowing us to cure most infected people and this stops the liver becoming damaged. Hepatitis C is common in Pakistan and the government is planning a massive national program to find and treat everyone who is infected. The government funded treatment program will fund therapy and assumes that the drugs will cure the vast majority of infected people and hence, in line with international recommendations they are not planning to evaluate treatment outcomes. The efficacy of the drugs used in Pakistan (sofosbuvir plus daclatasvir) have not been widely assessed in the Pakistani population and their efficacy is not yet proven. We therefore do not yet know how effective the drugs that will be used in Pakistan will be and we will study this by testing people after treatment to determine treatment effectiveness. This approach has been welcomed by the Pakistani government who recognise the importance of the data that we will generate from this observational study.

We will additionally look at the impact of hepatitis C on an individual's quality of life and how much they spend on healthcare by using questionnaires administered by the trial team.

We will look at viral factors influencing treatment failure by studying viral resistance by sequencing the virus from people who do and do not respond to treatment.

To determine whether or not re-infection is a significant problem in Pakistan we will look at people who have been cured of hepatitis C and retest them one year later. We will also retest people who initially tested negative to determine the annual infection rates in previously uninfected people. To determine risk factors for infection reinfected people and some of the non-reinfected cohort will be asked to complete a questionnaire on risk factors for infection.

One of the major effects of hepatitis C is induction of liver cancer. We will look at people who did and did not develop liver cancer following hepatitis C infection and we will compare viral sequences to see if there are viral variants that predispose to liver cancer.

This work will help make treatments more effective in Pakistan and we will work out, by modelling, how many people need to be cured to stop the spread of infection. We will look at which viruses cause cancer to help find better ways to screen and treat hepatitis C induced cancers.

In addition to this work, we will join colleagues in Pakistan to run a separate clinical trial of different treatments in people who did not respond to antiviral therapy. It is noted here to ensure that the comprehensive nature of this research study is recognised.

The study procedure will include:

* To screen, informed written consent will be obtained from participants who fulfil the inclusion eligibility criteria. This will consist of any person in the community over 18 years of age.
* Data will be collected on paper CRFs which will be securely stored prior to the data being transferred to a secure on-line database. Paper records will be retained as primary source documents.
* A screening log will be completed which will record the age group, gender and brief details of eligibility or ineligibility as well as administration errors and reasons why the patient may not have been willing to participate.
* After obtaining written informed consent, a study specific participant identification number (ID) will be assigned to the participant.
* Initial HCV screening of individuals will be with a rapid HCV antibody test (SD Rapid Test 02FK10, Standard Diagnostics, Inc., Republic of Korea) which is a WHO pre-qualified test and has been validated previously at AKU. The output on the RDT cassette is read independently by two observers (who are trained and certified) and recorded accordingly. Discrepant RDT results will be resolved with HCV RNA testing.
* In people who are HCV antibody positive 10ml blood will be collected for HCV RNA testing, CBC, AST, ALT, serum creatinine and HBsAg.
* For patients who are HCV RNA positive and who enter the study before commencing treatment, prior to therapy (Day 1) the patient will be asked to complete:
* Demographic and risk factor questions
* QOL EQ5D-3L questionnaire
* Productivity questionnaire
* Healthcare usage questionnaire
* This will be completed by all patients until 200 HCV positive and 1000 HCV patients as well as 50 cirrhotic patients are identified.
* The presence of cirrhosis will be determined using a non-invasive test for fibrosis such as the APRI using cut-offs of < 1.5, as well as Fibroscan where available. Patients who have liver cirrhosis demonstrated by high APRI or a fibro scan or ultrasound or a liver biopsy if available will be treated for 24 weeks (6 months). Patients who do not demonstrate liver cirrhosis will be treated with a course of 12 weeks (three months) as per the standard regimen.
* Patients on their first clinic visit will have a thorough medical history taken with a general and a systemic physical examination, HCV status will be relayed to the patient and counselling regarding the disease and treatment will be untaken where needed.
* Patients will undergo government/NGO or self-funded sofosbuvir + daclatasvir first-line treatment.
* A blood sample will be taken 12 weeks (range 10-18 weeks) after the completion of treatment regimen for SVR testing.
* HCV negative individual will be recalled for repeat HCV antibody testing after 12 months (range 11-14 months). They will be asked to complete risk factor questions if they are newly HCV antibody positive. Additionally, 4 times as many matched HCV negative individuals will also complete the risk factor questionnaire.
* Those who were HCV positive at screening and have successful first-line treatment will be invited 12 months after the completion of the treatment regimen for repeat HCV testing by HCV core antigen. All re-infected patients will also undertake:
* Risk factor questions
* QOL EQ5D-3L questionnaire
* Productivity questionnaire
* Blood sample for viral sequencing
* Four times as many HCV negative matched individuals will also complete the three questionnaires.
* Cost effectiveness of the treatment regimen will be measured from the Pakistan health service perspective. Costings for the drugs, clinic, laboratory testing, staff and facility costs associated with each treatment regimen per patient will be calculated.
* Patients will be monitored monthly, and treatment will be discontinued if they develop cirrhosis/decompensated liver disease. If the patient becomes pregnant or starts nursing an infant. Patients will also stop treatment if they develop major side effects or major weight loss.
* Participants may withdraw from a research study for any reason, without penalty. For evaluation and reporting purposes, researchers may ask participants for their reasons for early withdrawal.

Laboratory tests during the trial will include:

1. Blood tests taken to measure:

   * HCV RNA testing
   * HCV core antigen testing
   * Hepatitis B serum antigen
   * Serum asparate aminotransferase (AST)
   * Serum alanine aminotransferase (ALT)
   * Serum albumin
   * AST/ALT ratio
   * Platelet count
   * APRI [(AST/AST upper limit))/platelet count] x100
   * Alpha-fetopotein (AFP)
   * Total bilirubin
   * Serum Creatinine
   * Sodium
   * Prothrombin time (PT)/ International normalized ratio (INR)
2. Model for end of stage liver disease (MELD) score
3. Fibroscan or liver biopsy to assess cirrhosis
4. Blood sample to measure sustained virological response (SVR - defined as HCV RNA undetectable using a molecular diagnostic assay with a sensitivity of <100 IU/ml) 12 weeks after the completion of the second-line antiviral therapy. Once all participants have their SVR assess this will be the end of the study.

HCV whole genome sequencing to detect viral polymorphisms associated with treatment outcome:

* For all treatment failure patients, the stored baseline plasma samples will be used for nucleic acid extraction. NGS library preparation will be performed and HCV whole genome sequences will be generated.
* Baseline plasma samples from the same number of patients who have achieved SVR and are matched according to age, sex, cirrhosis and HCV infection risk factors will also be used to generate HCV whole genome sequences.
* We will use logistic regression to test for association between all polymorphic sites in the virus polyprotein and treatment outcome accounting for confounding factors.

HCV whole genome sequencing to detect viral polymorphisms associated with HCC:

* For all the patients enrolled in the HCC study (patients with HCV associated HCC), stored baseline plasma samples will be used for nucleic acid extraction. NGS library preparation will be performed and HCV whole genome sequences will be generated.
* Baseline plasma samples from the same number of patients with HCV associated cirrhosis which are matched according to age, sex and HCV infection risk factors will also be used to generate HCV whole genome sequences. These patients will be chosen from the ~5000 enrolled in the treatment study.
* We will use logistic regression to test for association between all polymorphic sites in the virus polyprotein and HCC accounting for confounding factors. Additionally, we will run a focused analysis on NS5B A150V polymorphism and other viral polymorphism associated with HCC

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18yrs old
* Willing to undergo hepatitis C testing
* Able and willing to give informed consent
* Willing to return in 12 months time for repeat testing
* Resident in area and not planning to leave the region

Exclusion Criteria:

* Unwilling to give consent
* Unwilling or unable to undergo the necessary procedures
* Clinically significant illness (other than HCV) or other major medical condition that may interfere with the subject's treatment, assessment or compliance with protocol.
* Co-morbidities limiting life expectancy to less than 12 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment of uninfected and infected people will be from two provinces in Pakistan (Sindh and Punjab) where there is a high prevalence of HCV. Recruitment will reflect the community sample.
Sampling Method: Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
SVR | 12 weeks after treatment completion
  After first-line treatment, SVR will be measured to record treatment failure or success
Incidence of new infections | 12 months after screening
  Measure HCV antibodies in people who initially tested HCV antibody negative at screening.
Incidence of re-infection | 12 months after first SVR test.
  In patients who achieved an SVR after first-line treatment will then be tested for HCV core antigen over 12 months.

SECONDARY OUTCOMES:
Health related Quality of Life | Screening stage
  Determined by an EQ-5D-3L questionnaire in 200 HCV positives and at least 1000 negatives and 50 cirrhotic patients
Health care costs and productivity assessment associated with HCV infection | screening stage
  Questionnaires in 200 HCV positives and at least 1000
Risk assessment | 12 months
  Assess risk factors using questionnaires for HCV infection in 200 HCV positives and at least 1000. Then after 12months in HCV negatives
Viral polymorphisms in HCV | 2 years
  Investigating the frequencies in people who respond to therapy compared with those who do not achieve SVR Identified using whole viral genome sequencing in all patients who do not respond to therapy and age, gender and liver disease matched controls
Viral polymorphisms in HCV associated with hepatocellular carcinoma | 4 years
  Identify using whole viral genome sequencing and polymorphism frequencies in 400 people with HCV associated liver cirrhosis without liver cancer compared with 400 people who do have liver cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Graham R Foster, MBBS, Principal Investigator — Queen Mary University
Locations (1):
- Aga Khan University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] El-Akel W, El-Sayed MH, El Kassas M, El-Serafy M, Khairy M, Elsaeed K, Kabil K, Hassany M, Shawky A, Yosry A, Shaker MK, ElShazly Y, Waked I, Esmat G, Doss W. National treatment programme of hepatitis C in Egypt: Hepatitis C virus model of care. J Viral Hepat. 2017 Apr;24(4):262-267. doi: 10.1111/jvh.12668. Epub 2017 Feb 1. PMID 28145032
- [Result] Smith D, Magri A, Bonsall D, Ip CLC, Trebes A, Brown A, Piazza P, Bowden R, Nguyen D, Ansari MA, Simmonds P, Barnes E; STOP-HCV Consortium. Resistance analysis of genotype 3 hepatitis C virus indicates subtypes inherently resistant to nonstructural protein 5A inhibitors. Hepatology. 2019 May;69(5):1861-1872. doi: 10.1002/hep.29837. Epub 2018 Apr 27. PMID 29425396
- [Result] Zeuzem S, Foster GR, Wang S, Asatryan A, Gane E, Feld JJ, Asselah T, Bourliere M, Ruane PJ, Wedemeyer H, Pol S, Flisiak R, Poordad F, Chuang WL, Stedman CA, Flamm S, Kwo P, Dore GJ, Sepulveda-Arzola G, Roberts SK, Soto-Malave R, Kaita K, Puoti M, Vierling J, Tam E, Vargas HE, Bruck R, Fuster F, Paik SW, Felizarta F, Kort J, Fu B, Liu R, Ng TI, Pilot-Matias T, Lin CW, Trinh R, Mensa FJ. Glecaprevir-Pibrentasvir for 8 or 12 Weeks in HCV Genotype 1 or 3 Infection. N Engl J Med. 2018 Jan 25;378(4):354-369. doi: 10.1056/NEJMoa1702417. PMID 29365309
- [Result] Lim AG, Walker JG, Mafirakureva N, Khalid GG, Qureshi H, Mahmood H, Trickey A, Fraser H, Aslam K, Falq G, Fortas C, Zahid H, Naveed A, Auat R, Saeed Q, Davies CF, Mukandavire C, Glass N, Maman D, Martin NK, Hickman M, May MT, Hamid S, Loarec A, Averhoff F, Vickerman P. Effects and cost of different strategies to eliminate hepatitis C virus transmission in Pakistan: a modelling analysis. Lancet Glob Health. 2020 Mar;8(3):e440-e450. doi: 10.1016/S2214-109X(20)30003-6. PMID 32087176
- [Result] Foster GR, Afdhal N, Roberts SK, Brau N, Gane EJ, Pianko S, Lawitz E, Thompson A, Shiffman ML, Cooper C, Towner WJ, Conway B, Ruane P, Bourliere M, Asselah T, Berg T, Zeuzem S, Rosenberg W, Agarwal K, Stedman CA, Mo H, Dvory-Sobol H, Han L, Wang J, McNally J, Osinusi A, Brainard DM, McHutchison JG, Mazzotta F, Tran TT, Gordon SC, Patel K, Reau N, Mangia A, Sulkowski M; ASTRAL-2 Investigators; ASTRAL-3 Investigators. Sofosbuvir and Velpatasvir for HCV Genotype 2 and 3 Infection. N Engl J Med. 2015 Dec 31;373(27):2608-17. doi: 10.1056/NEJMoa1512612. Epub 2015 Nov 17. PMID 26575258
- [Result] Wing PAC, Jones M, Cheung M, DaSilva S, Bamford C, Jason Lee WY, Aranday-Cortes E, Da Silva Filipe A, McLauchlan J, Smith D, Irving W, Cunningham M, Ansari A, Barnes E, Foster GR. Amino Acid Substitutions in Genotype 3a Hepatitis C Virus Polymerase Protein Affect Responses to Sofosbuvir. Gastroenterology. 2019 Sep;157(3):692-704.e9. doi: 10.1053/j.gastro.2019.05.007. Epub 2019 May 10. PMID 31078622
- [Result] Huang R, Rao H, Xie Q, Gao Z, Li W, Jiang D, Mo H, Massetto B, Stamm LM, Brainard DM, Wei L. Comparison of the efficacy of sofosbuvir plus ribavirin in Chinese patients with genotype 3a or 3b HCV infection. J Med Virol. 2019 Jul;91(7):1313-1318. doi: 10.1002/jmv.25454. Epub 2019 Apr 3. PMID 30861150
- [Result] Lim AG, Qureshi H, Mahmood H, Hamid S, Davies CF, Trickey A, Glass N, Saeed Q, Fraser H, Walker JG, Mukandavire C, Hickman M, Martin NK, May MT, Averhoff F, Vickerman P. Curbing the hepatitis C virus epidemic in Pakistan: the impact of scaling up treatment and prevention for achieving elimination. Int J Epidemiol. 2018 Apr 1;47(2):550-560. doi: 10.1093/ije/dyx270. PMID 29309592
- [Derived] Arif A, Hasnain A, Chaudhry A, Asim M, Shafqat MN, Altaf A, Saba N, Kemos P, Ansari MA, Barnes E, Metcalfe C, Vickerman P, Qureshi H, Hamid S, Choudhry AA, Niaz SK, Foster GR, Choudhry N. HepFREEPak: protocol for a multi-centre, prospective observational study examining efficacy and impact of current therapies for the treatment of hepatitis C in Pakistan and reporting resistance to antiviral drugs: study protocol. BMC Public Health. 2023 Dec 18;23(1):2529. doi: 10.1186/s12889-023-17290-3. PMID 38110885

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT04943588/SAP_000.pdf